CLINICAL TRIAL: NCT07217015
Title: A Phase 2b, Randomized, Double-blind, Placebo-controlled, Parallel-group, Multicenter, Dose-ranging Study With an Open-label Period Investigating the Efficacy and Safety Profile of KT-621 Administered Orally to Participants With Moderate to Severe Atopic Dermatitis
Brief Title: A Study of KT-621 Administered Orally to Participants With Moderate to Severe Atopic Dermatitis
Acronym: BROADEN2
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: Kymera Therapeutics, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Triple | Purpose: Treatment
Other Study IDs: KT621-AD-201; 2025-522370-36-00 (EU CTIS Number)
Record Dates: First submitted 2025-10-13; First posted 2025-10-15 (Actual); Last update posted 2026-01-14 (Actual); Status verified 2026-01

CONDITIONS: Atopic Dermatitis
Keywords: STAT6; stat6 degrader; targeted protein degrader; Phase 2; Phase 2b; kt-621
MeSH Terms: conditions — Dermatitis, Atopic

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (4):
- Group 1: KT-621 Dose 1 (Experimental)
  Interventions: Drug: KT-621
- Group 2: KT-621 Dose 2 (Experimental)
  Interventions: Drug: KT-621
- Group 3: KT-621 Dose 3 (Experimental)
  Interventions: Drug: KT-621
- Group 4: Placebo (Placebo Comparator)
  Interventions: Other: Placebo

INTERVENTIONS:
Drug: KT-621 — Oral drug
  Arms: Group 1: KT-621 Dose 1; Group 2: KT-621 Dose 2; Group 3: KT-621 Dose 3
Other: Placebo — Oral placebo matched to KT-621
  Arms: Group 4: Placebo

SUMMARY:
This phase 2b study is designed to evaluate the safety and efficacy of KT-621 in adult and adolescent participants with moderate-to-severe atopic dermatitis (AD), a common form of eczema. The main goals of this study are to learn how effective KT-621 is at reducing the severity and extent of AD, the safety and tolerability of KT-621, how KT-621 behaves in the body, and how the body responds to KT-621. This is a 16-week double-blind, placebo-controlled study with a 52-week open-label period.

ELIGIBILITY:
Inclusion Criteria:

* Must be 12 to 75 years of age, inclusive, at the time of signing the IAF (informed assent form) and/or ICF (informed consent form).
* Must have chronic AD that has been present for at least 3 years before the Screening visit.
* Must have an EASI score ≥ 16 at the Screening and Baseline visits.
* Must have a vIGA-AD score ≥ 3 (scale of 0 to 4) at the Screening and Baseline visits.
* Must have at least 10% BSA of AD involvement at the Screening and Baseline visits.
* Must have a weekly average Peak Pruritus NRS value ≥ 4 at the Baseline visit.
* Must have a documented history within the 6 months prior to the Baseline visit of either an inadequate response to, or inability to take, topical medications for the treatment of AD.
* Must apply a stable dose of moisturizer at least twice daily for at least 7 consecutive days immediately prior to the Baseline visit. Participants should be willing to continue using moisturizer twice daily during the study.
* Must be willing and able to comply with scheduled visits, treatment plan, laboratory tests, other study-related procedures, and questionnaires, including completing the electronic diary (e-diary), for the duration of the study as required by the study protocol.
* Must agree to contraceptive requirements in compliance with the clinical study and local requirements.

Exclusion Criteria:

* Must not have an unstable course of AD (spontaneously improving or rapidly deteriorating) as determined by the Investigator in the 4 weeks before the baseline visit.
* Must not have other skin conditions, such as contact dermatitis, psoriasis, tinea corporis, or lupus erythematosus, that may interfere with study assessments.
* Must not have a clinically relevant history of respiratory, gastrointestinal (GI), renal, hepatic, hematological, lymphatic, endocrinological, neurological, cardiovascular, psychiatric, musculoskeletal, genitourinary, immunological, ophthalmological, or connective tissue diseases or disorders.
* Must not have any surgical or medical procedure planned during participation in the study.
* Must not have a history of alcohol or substance abuse within the previous 2 years.
* Must not be pregnant or breastfeeding; must not be a woman planning to become pregnant or breastfeed during the study.
* Must not have a history of lack of response to any medication targeting interleukin (IL)-4, IL-13, and/or janus kinase (JAK)- signal transducer and activator of transcription (STAT) pathways (e.g. dupilumab, tralokinumab, upadacitinib, abrocitinib) at approved doses after at least 16 weeks of therapy.
* Must not have results from clinical laboratory safety tests that are outside the local reference range at Screening.
* Must not have been dosed with any investigational drug or device in a clinical study within 8 weeks or 5 half-lives (whichever is longer) of KT-621 administration.
* Female participants of childbearing potential must not have a positive or undetermined pregnancy result at the Screening and baseline visits.
* Must not have any known factor, condition, or disease that might interfere with treatment compliance, study conduct or interpretation of the results.
* Must not be taking or have taken any prespecified prohibited therapies within a specific timeframe as evaluated by the Investigator.
* Must not have a known sensitivity to any of the components of KT-621.
* Must not be a member of the investigational team or his/her immediate family.

Ages: 12 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult, Older Adult
Enrollment: 200 (Estimated)
Dates: Start 2025-11-24 (Actual); Primary Completion 2027-06 (Estimated); Study Completion 2028-06 (Estimated)

PRIMARY OUTCOMES:
Change from baseline in Eczema Area and Severity Index (EASI) score | From baseline through Week 16

SECONDARY OUTCOMES:
Incidence of treatment-emergent adverse events (TEAEs) | From baseline through Week 16, and from Week 16 through Week 68
Incidence of treatment-emergent serious adverse events (SAEs) | From baseline through Week 16, and from Week 16 through Week 68
Percentage change from baseline in body surface area (BSA) affected by AD | From baseline to Week 16 and to Week 68
Percentage change from baseline in the Peak Pruritus NRS score | From baseline to Week 16, and to Week 68
Proportion of participants with at least a 4-point improvement from baseline in the Peak Pruritus Numerical Rating Scale (NRS) | At Week 16 and at Week 68
Proportion of participants who achieve a validated Investigator Global Assessment Scale for Atopic Dermatitis (vIGA-AD) score of 0 to 1 (on a 5-point scale) and a reduction from the baseline value of at least 2 points | At Week 16 and at Week 68
Proportion of participants with EASI-50, EASI-75, and EASI-90 | At Week 16 and at Week 68
Percentage change from baseline in the EASI score | From baseline to Week 68
Percentage change from baseline in the SCORing Atopic Dermatitis (SCORAD) score | From baseline to Week 16, and to Week 68
Change from baseline in the Patient-Oriented Eczema Measure (POEM) | From baseline to Week 16, and to Week 68
Change from baseline in the Dermatology Life Quality Index (DLQI) or the Children's Dermatology Life Quality Index (c-DLQI) | From baseline to Week 16, and to Week 68
Plasma concentration of KT-621 derived from plasma concentration time data | From baseline to Week 16, and to Week 68

CONTACTS AND LOCATIONS:
Locations (19):
- United States (11):
  - Kymera Investigative Site, Birmingham, Alabama
  - Kymera Investigative Site, North Little Rock, Arkansas
  - Kymera Investigative Site, Los Angeles, California
  - Kymera Investigative Site, Santa Monica, California
  - Kymera Investigative Site, Delray Beach, Florida
  - Kymera Investigative Site, Miami, Florida
  - Kymera Investigative Site, Miramar, Florida
  - Kymera Investigative Site, Ann Arbor, Michigan
  - Kymera Investigative Site, Fargo, North Dakota
  - Kymera Investigative Site, Philadelphia, Pennsylvania
  - Kymera Investigative Site, San Antonio, Texas
- Australia (3):
  - Kymera Investigative Site, Darlinghurst, New South Wales
  - Kymera Investigative Site, Brisbane, Queensland
  - Kymera Investigative Site, Melbourne, Victoria
- Canada (5):
  - Kymera Investigative Site, Kelowna, British Columbia
  - Kymera Investigative Site, Surrey, British Columbia
  - Kymera Investigative Site, Markham, Ontario
  - Kymera Investigative Site, Ottawa, Ontario
  - Kymera Investigative Site, Toronto, Ontario

IPD SHARING:
Plan to Share IPD: No